CLINICAL TRIAL: NCT03523052
Title: The Chinese Parkinson's Disease With SNCA Variants Registry
Brief Title: Chinese PD-SNCA Registry
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CPD-SNCAR
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese PD-SNCA Registry(CPD-SNCAR) is to develop a database of patients of Parkinson's disease with a-synuclein (SNCA) gene variants in mainland China.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common disorder among neurodegenerative diseases. SNCA is the first gene implicated in monogenic parkinsonism. However, some polymorphisms of SNCA gene such as rs894278 and rs11931074 can affect the risk of sporadic PD. The investigators aim to establish a database of PD with SNCA variants and characterize the clinical manifestation of these patients in mainland China.

Method:

1. Peripheral blood from patients has been tested to have SNCA gene variants.
2. Clinical manifestation will be measured by scales and neurological tests. Standard scales include: Unified Parkinson's Disease Rating Scale(UPDRS), Hoehn-Yahr stages, Non-Motor Symptoms Scale (NMSS), mini-mental state examination (MMSE), Parkinson disease sleep scales (PDSS), Rapid Eye Movement Sleep Behaviour Disorder Questionnaire(RBDQ-HK), Epworth Sleepiness Scale (ESS), Rome III functional constipation scale, the Scale for Outcomes in PD for Autonomic Symptoms (SCOPA-AUT), Parkinson Fatigue Scale (PFS), Cambridge-Hopkins Restless Legs Syndrome questionnaire (CHRLSq), Hyposmia rating scale(HRS), Hamilton depression scale, the 39-item Parkinson's Disease Questionnaire(PDQ-39), Freezing of gait scale(FOG), dyskinesia related scales, Wearing-off scale(WO).
3. The investigators will also exam the blood biomarkers of PD such as uric acid and peripheral inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD by the United Kingdom Parkinson's Disease Society Brain Bank clinical diagnostic criteria or other standard criteria; PD patients detected with positive SNCA variants

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PD patients with SNCA variants
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Database of Parkinson's disease with SNCA variants | 10 years
  Establish the database of Parkinson's disease with SNCA variants in mainland China.
Clinical feature | 10 years
  Characterize the clinical feature in patients of Parkinson's disease with SNCA variants

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Result] Hu Y, Tang B, Guo J, Wu X, Sun Q, Shi C, Hu L, Wang C, Wang L, Tan L, Shen L, Yan X, Zhang H. Variant in the 3' region of SNCA associated with Parkinson's disease and serum alpha-synuclein levels. J Neurol. 2012 Mar;259(3):497-504. doi: 10.1007/s00415-011-6209-4. Epub 2011 Aug 19. PMID 21853288
- [Result] Ai SX, Xu Q, Hu YC, Song CY, Guo JF, Shen L, Wang CR, Yu RL, Yan XX, Tang BS. Hypomethylation of SNCA in blood of patients with sporadic Parkinson's disease. J Neurol Sci. 2014 Feb 15;337(1-2):123-8. doi: 10.1016/j.jns.2013.11.033. Epub 2013 Dec 1. PMID 24326201
- [Result] Guo JF, Li K, Yu RL, Sun QY, Wang L, Yao LY, Hu YC, Lv ZY, Luo LZ, Shen L, Jiang H, Yan XX, Pan Q, Xia K, Tang BS. Polygenic determinants of Parkinson's disease in a Chinese population. Neurobiol Aging. 2015 Apr;36(4):1765.e1-1765.e6. doi: 10.1016/j.neurobiolaging.2014.12.030. Epub 2015 Jan 6. PMID 25623333
- [Result] Wei Y, Yang N, Xu Q, Sun Q, Guo J, Li K, Liu Z, Yan X, Zhu X, Tang B. The rs3756063 polymorphism is associated with SNCA methylation in the Chinese Han population. J Neurol Sci. 2016 Aug 15;367:11-4. doi: 10.1016/j.jns.2016.05.037. Epub 2016 May 19. PMID 27423554